CLINICAL TRIAL: NCT02217657
Title: "Bidirectional Conduction Block of Left Atrial Anterior Line in Patients With Left Atrial Ablation - Reduction of RF Applications Using the Thermocool SmartTouch Contact Force Sensing Catheter
Brief Title: SmartTouch Catheter for Left Anterior Line - SmarT Line Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Heidi Estner, Director Interventional Electrophysiology, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MucM001-13
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Smart-Touch; Contact force
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- operator informed to contact force (Active Comparator): Thermocool Smart Touch Catheter, operator informed to contact force (Biosense Webster)
  Interventions: Device: Thermocool Smart Touch Catheter
- operator blinded to contact force (Experimental): Thermocool Smart Touch catheter, operator blinded to contact force information (Biosense Webster)
  Interventions: Device: Thermocool Smart Touch Catheter

INTERVENTIONS:
Device: Thermocool Smart Touch Catheter — Physician informed to contact force

SUMMARY:
This prospective, randomized study will investigate, if information of the catheter force during ablation of a left anterior line does reduce total RF application time by prevention of ineffective lesions.

DETAILED DESCRIPTION:
Catheter ablation has emerged as a realistic therapeutic option for symptomatic atrial fibrillation (AF).

The three main techniques described for ablation of persistent AF include pulmonary vein (PV) isolation, ablation based on electrogram analysis, and left atrial (LA) linear lesions.

The ideal endpoint of linear lesions should be complete electrical block; however, this is technically challenging, time consuming, and potentially hazardous. The ST catheter combined with 3D mapping and navigation software, gives physicians a real-time, objective measure of tip-to-tissue contact force during the catheter ablation procedure and will allow physicians to more safely and effectively treat atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic atrial fibrillation and additional substrate modification or perimitral flutter
* Patients with persistent atrial fibrillation
* Patients with perimitral flutter
* Patients with recurrence after a circumferential PV isolation procedure
* Patients with paroxysmal atrial fibrillation and AF episodes lasting > 7 days
* Patients (>18 und <80 Jahre)

Exclusion Criteria:

* moderate to severe valvular heart disease,
* congenital heart disease
* reduced left ventricular function (ejection fraction <35%)
* any reversible cause for atrial fibrillation (e.g. hyperthyroidism)
* intracardiac thrombi documented by transesophageal echocardiography
* myocardial infarction within 3 months, cardiac surgery in the previous three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Duration of total RF application until bidirectional conduction block across the anterior line is achieved (including a waiting period of 30 minutes) | 30 minutes

SECONDARY OUTCOMES:
Achievement of primary endpoint (bidirectional conduction block at an anterior line) | 6 months
  Achievement of primary endpoint (bidirectional conduction block at an anterior line). Procedure Duration. Reduction of local potential amplitude during SR or atrial fibrillation after 60 seconds of ablation. Freedom of any atrial tachyarrhythmia at 7 day holter 3 and 6 months after a single ablation procedure. Freedom of any symptoms of atrial arrhythmias 6 months after ablation (except during blanking period of 6 weeks). Confirmation of gap-freeness in MRI (3-6 months after ablation). Quality of Life (atrial fibrillation symptom checklist und major depression index) pre, 3 and 6 months after Ablation. Safety (bleeding, pericardial effusion, thrombembolic events).

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Estner, MD, Principal Investigator — Munich University Clinic, Campus Großhadern
Locations (1):
- Munich University Clinic, Campus Großhadern, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fichtner S, Wakili R, Rizas K, Siebermair J, Sinner MF, Wiktor T, Lackermair K, Schuessler F, Olesch L, Rainer S, Kaab S, Curta A, Kramer H, Estner HL. Benefit of Contact Force Sensing Catheter Technology for Successful Left Atrial Anterior Line Formation: A Prospective Randomized Trial. Biomed Res Int. 2018 Sep 18;2018:9784259. doi: 10.1155/2018/9784259. eCollection 2018. PMID 30320138